CLINICAL TRIAL: NCT03086811
Title: "Improved Mother Infant Feeding Interaction (MI-FI) at 12 Months With Very Early Parent
Brief Title: "Improved Mother Infant Feeding Interaction (MI-FI) at 12 Months With Very Early Parent Training"
Acronym: MI-FI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0156-11-RMB
Record Dates: First submitted 2017-03-16; First posted 2017-03-22 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Picky Eaters, Feeding Interaction, Good Enough Parenting, Family Meals, Emotional Eating Prevention
Keywords: feeding interaction, infant eating habits, hunger satiety cues, childhood obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Intervention group got 4 sequential weekly training meetings, in small workshop groups setting, by a highly experience pediatric dietitian and social worker. The program covered nutritional aspects, as well as feeding and parenting topics. Training took place when infants were 4-6 months old. Thereafter, internet-based support continued until infants reached 12 months. The control group received customary support via municipal mother-child health clinics. Mealtime interactions by videotaped home setting feeding were documented at 12-13 months.
Who Masked: Outcomes Assessor
Masking Description: Mealtime interactions by videotaped home setting feeding were evaluated using the Chatoor feeding scale by blinded to group viewers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): First time mothers, when infants were ages 4-6 months old, took part in a training program in small group setting (10-12 mother-infants). the program continued for a month, with 4 weekly meetings. group coordinators were a highly experienced pediatric dietitian, and a social worker. Training topics addressed were infant healthy nutrition and growth, feeding skills, obesity and emotional feeding prevention, parenting. Thereafter, mothers were encouraged to stay in contact with the trainers, till infants reached age 12 months and data was collected using video taping of mealtime feeding interactions at home setting environment. Mother Infant Feeding Interaction very early training
  Interventions: Behavioral: Mother Infant Feeding Interaction very early training
- control group (No Intervention): Control group first time mothers were recruited when infants were around 11-12 months of age for data collection of mealtime feeding interactions taping at home setting environment. They received during this year the official support and training given in municipality care centers.

INTERVENTIONS:
Behavioral: Mother Infant Feeding Interaction very early training — weekly training meetings on 4 topics:
  1. What - proper nutrition and supplements for solid feeding phase (dietitian); What - the meaning of feeding to mother and infant (social worker).
  2. Who - feeding skills - knowledge and actual practices
  3. From anxiety to serenity - knowledge concerning growth patterns and common physical and emotional issues troubling parents of infants 4-12 months old.
  4. Prevention of obesity and emotional eating - practical advise and tips.
  Arms: intervention group

SUMMARY:
Rise in childhood obesity and poor eating habits and eating problems is apparent over the last decades. Parents are at lose what the correct way to tackle these problems may be. This study examined whether professional behavioral and nutritional training of first time mothers improves feeding relationship and infants eating habits at 12 months.

DETAILED DESCRIPTION:
From 166 first time mother-infant recruited, 128 completed the trail. Intervention group, mother-infant dyads got a month long weekly based training in small workshop groups about nutrition, feeding and parenting when infants were 4-6 months old. training was given by a highly experience pediatric dietitian and social worker. Thereafter, internet-based support continued until infants reached 12 months. The control group received customary support via municipal mother-child health clinics. Mealtime interactions were videotaped at home setting at 12 months and were evaluated using the Chatoor feeding scale by blinded (to group) viewers.

ELIGIBILITY:
Inclusion Criteria:

* normal and healthy pregnancy
* full term delivery of infants
* infants with a normal birth weight and no health problems
* Mothers recruited had at least a high school education
* mothers lived near to or in the city (important for video taping)

Exclusion Criteria:

* Mothers with mental illness in the present or the past (such as schizophrenia, depression or an eating disorder)
* infants with chronic diseases that required specific diets (such as milk allergy) or gastrointestinal diseases (celiac disease, type 1 diabetes, Crohn's disease etc.)

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 166 (Actual)
Dates: Start 2011-10-25 (Actual); Primary Completion 2013-07-21 (Actual); Study Completion 2013-07-21 (Actual)

PRIMARY OUTCOMES:
Chatoor feeding scale | 12 months
  the Chatoor observational scale for Mother-Infant interaction during feeding was purchased from the Chatoor Center. The Scale consists of 46 mother and infant behavior modes which are rated throughout the feeding session. Five subscale scores are derived: 1) Dyadic Reciprocity, 2) Dyadic Conflict, 3) Talk and Distraction, 4) Struggle for Control, and 5) Maternal Non-Contingency. The CFS has been demonstrated to discriminate between infants with and without feeding disorders and can be used with infants and toddlers ranging from 1 month to 3 years of age (Chatoor et al, 1997).

SECONDARY OUTCOMES:
eating habitts | 12 months
  Self reported questionnaires of Golan et al checking eating habits and obesogenic environment at home

CONTACTS AND LOCATIONS:
Overall Officials: Ron Shaoul, MD, Principal Investigator — Pediatric Gastroenterology Unit, Ruth Rappaport Children's Hospital Rambam Health Care Campus, Haifa, Israel, Rappaport Faculty of Medicine;

IPD SHARING:
Plan to Share IPD: Undecided
The investigators plan to publish results of the research project in peer reviewed journals. However, individual data collected, such as video taping of family meals will not be shared.

REFERENCES:
- [Background] Redsell SA, Edmonds B, Swift JA, Siriwardena AN, Weng S, Nathan D, Glazebrook C. Systematic review of randomised controlled trials of interventions that aim to reduce the risk, either directly or indirectly, of overweight and obesity in infancy and early childhood. Matern Child Nutr. 2016 Jan;12(1):24-38. doi: 10.1111/mcn.12184. Epub 2015 Apr 20. PMID 25894857
- [Background] Bryant-Waugh R, Markham L, Kreipe RE, Walsh BT. Feeding and eating disorders in childhood. Int J Eat Disord. 2010 Mar;43(2):98-111. doi: 10.1002/eat.20795. PMID 20063374
- [Background] Meadows N. Assessment and management of feeding difficulties in infants. Community Pract. 2015 Feb;88(2):45-7. No abstract available. PMID 25720215
- [Background] Ammaniti M, Lucarelli L, Cimino S, D'Olimpio F, Chatoor I. Feeding disorders of infancy: a longitudinal study to middle childhood. Int J Eat Disord. 2012 Mar;45(2):272-80. doi: 10.1002/eat.20925. Epub 2011 Apr 14. PMID 21495054